CLINICAL TRIAL: NCT03864419
Title: A Phase I Study of Subcutaneous Rituximab Hyaluronidase Combined With Local Standard-of-Care Chemotherapy for the Treatment of Burkitt Lymphoma, Diffuse Large B-Cell Lymphoma or as Monotherapy for Kaposi Sarcoma Herpesvirus Associated Multicentric Castleman Disease in Pediatrics and Adults in Uganda
Brief Title: Rituximab Hyaluronidase in Combination With Chemotherapy in Treating Aggressive B-cell Lymphoma in Uganda
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed per SRC Low Accrual Policy
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1001799; U028 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2019-01493 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10040 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Burkitt Lymphoma; KSHV-associated Multicentric Castleman Disease; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Multi-centric Castleman's Disease; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Hyaluronoglucosaminidase; Cyclophosphamide; Vincristine; Methotrexate; Doxorubicin; Prednisone; deltacortene; Etoposide; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort I (pediatric BL) (Experimental): Patients receive cyclophosphamide IV and vincristine IV on day 1, and prednisone IV or PO on days 1-7 in the absence of disease progression or unacceptable toxicity. Patients then receive rituximab IV or rituximab hyaluronidase SC, cyclophosphamide IV, vincristine IV, and methotrexate IV on day 1. Cycles repeat every 14 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Rituximab and Hyaluronidase Human; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Methotrexate; Biological: Rituximab
- Cohort II (DLBCL) (Experimental): Patients receive rituximab IV or rituximab and hyaluronidase human SC, cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1, and prednisone PO on days 1-5 of cycle 1. Cycles repeat every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Rituximab and Hyaluronidase Human; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Drug: Etoposide; Biological: Rituximab
- Cohort III (Adult BL) (Experimental): Patients receive rituximab IV or rituximab and hyaluronidase human SC in day 1, etoposide IV, doxorubicin IV, and vincristine IV on days 1-4. Patients also receive cyclophosphamide IV on day 5 and prednisone PO on days 1-5. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Rituximab and Hyaluronidase Human; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Prednisone; Biological: Rituximab
- Cohort IV (MCD) (Experimental): Patients receive rituximab IV or rituximab and hyaluronidase human SC on days 1, 8, 15, and 22 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Rituximab and Hyaluronidase Human; Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab and Hyaluronidase Human — Given SC
  Other Names: Rituxan Hycela; Rituximab Plus Hyaluronidase; Rituximab/Hyaluronidase; Rituximab/Hyaluronidase Human
Drug: Cyclophosphamide — Given IV
  Other Names: Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal
  Arms: Cohort I (pediatric BL); Cohort II (DLBCL); Cohort III (Adult BL)
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine
  Arms: Cohort I (pediatric BL); Cohort II (DLBCL); Cohort III (Adult BL)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; Emthexat; Emtexate; Methotrexate LPF; Methylaminopterin; Methotrexatum
  Arms: Cohort I (pediatric BL)
Drug: Doxorubicin — Given IV
  Other Names: Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Cohort II (DLBCL); Cohort III (Adult BL)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: Adriamycine; Adriblastina; Doxolem; Doxorubicin.HCl
  Arms: Cohort II (DLBCL); Cohort III (Adult BL)
Drug: Prednisone — Given PO
  Other Names: Deltacortene; Decorton; Decortisyl; DeCortin; Deltacortisone; Econosone
  Arms: Cohort II (DLBCL); Cohort III (Adult BL)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Vepesid
  Arms: Cohort II (DLBCL)
Biological: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar JHL1101; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; RTXM83; Truxima

SUMMARY:
This phase I trial studies how well rituximab hyaluronidase and combination chemotherapy work in treating patients in Uganda with Burkitt lymphoma, diffuse large B-cell lymphoma, or Kaposi sarcoma herpesvirus associated multicentric Castleman disease. Rituximab hyaluronidase is a combination of rituximab and hyaluronidase. Rituximab binds to a molecule called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Hyaluronidase allows rituximab to be given by injection under the skin. Giving rituximab and hyaluronidase by injection under the skin is faster than giving rituximab alone by infusion into the blood. Drugs used in chemotherapy, such as cyclophosphamide, vincristine, methotrexate, etoposide, doxorubicin, and prednisone work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. While rituximab has a clear survival benefit in patients within developed countries, differences in supportive care and infectious co-morbidities require special attention. Giving rituximab hyaluronidase alone or in combination with chemotherapy may work better in treating patients with Burkitt lymphoma, diffuse large B-cell lymphoma, or Kaposi sarcoma herpesvirus associated multicentric Castleman disease compared to chemotherapy alone in Uganda.

DETAILED DESCRIPTION:
OUTLINE:

Open-label Phase I study characterizing the safety, tolerability, and activity of subcutaneous rituximab hyaluronidase (sqR) alone (KSHV-MCD), or combined with local standard of care chemotherapy (BL or DLBCL), in 2 age-based cohorts of patients:

1. Cohort 1: Age >= 15
2. Cohort 2: Age: 2-14

sqR dose for Cohort 1 (adults) will be 1400 mg (flat dose); sqR dose for Cohort 2 (pediatrics) will depend on patient weight: >= 35 kg: 1400 mg, < 35 kg: 700 mg. For all participants, sqR will be administered with local standard of care chemotherapy (BL, DLBCL) or alone (KSHV-MCD), and supportive care.

Each cohort comprises two Therapy Groups. Therapy Group 1: up to 6 participants and will receive the first cycle of rituximab IV, and subsequent cycles as flat-dose sqR. Therapy Group 2: up to 12 participants and will receive flat-dose sqR for all cycles.

Disease-specific chemotherapy to be administered with rituximab hyaluronidase include:

PEDIATRIC BURKITT LYMPHOMA (BL): cyclophosphamide, vincristine and prednisone followed by 6 cycles of cyclophosphamide, vincristine, and methotrexate (COP-COM).

DLBCL: 6 cycles of cyclophosphamide, doxorubicin, vincristine and prednisone PO on days 1-5 of cycle 1 (CHOP).

ADULT BL: 6 cycles modified dose: etoposide, doxorubicin, vincristine, cyclophosphamide and prednisone PO on days 1-5 (adjusted EPOCH).

KSHV-MCD: Rituximab or rituximab hyaluronidase SC on days 1, 8, 15, and 22.

After completion of study treatment, patients are followed up at 30 days, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histology and immunohistochemistry (CD20+) confirmed Burkitt lymphoma (BL), diffuse large B-cell lymphoma (DLBCL), or histology confirmed KSHV-associated multicentric Castleman disease with elevated blood KSHV viral load
* Cohort 1: Age should be equal to or greater than 15
* Cohort 2: Age: 2-15
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Able to provide informed consent (adults) or assent (children < 18 years) in English or Luganda
* Human immunodeficiency virus (HIV)-infected patients eligible if meet the following criteria:

  * CD4+ T-cell count > 200 cells/uL
  * HIV treatable with effective antiretroviral therapy that does not include agents with known significant drug-drug interactions with accompanying chemotherapy (ritonavir and cobicistat contraindicated)

Exclusion Criteria:

* Previous therapy for lymphoma or KSHV-multicentric Castleman disease (MCD)
* History of hypersensitivity to rituximab
* Pregnant or nursing women. Men or women may not participate unless they have agreed to use effective contraception during treatment and for 12 months following completion of therapy
* Inadequate organ function, unless attributed to lymphoma or KSHV-MCD
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 times upper limit of normal
* Creatinine > 2 times upper limit than normal or calculated creatinine clearance < 60 mL/min
* New York Heart Association (NYHA) cardiac failure class III or IV
* Patients with clinically significant anemia-hemoglobin less than 10 g/dL
* Central nervous system (CNS) masses consistent with lymphoma or untreated infection; leptomeningeal disease will not be excluded
* Patients with malignancy within 5 years, other than resected local skin cancer or limited Kaposi sarcoma (KS) (no known pulmonary KS)
* Patients with evidence of active infections including malaria and hepatitis B (participants with hepatitis B virus [HBV] controlled on antivirals will not be excluded)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 12 months
  Common Terminology Criteria for Adverse Events version 5.0 including unanticipated problems and grade 3-5 adverse events (AEs) at least probably related to subcutaneous rituximab hyaluronidase (sqR) administration.
Number of participants that result in sufficient pharmacodynamic criteria | Up to 12 months
  Pharmacodynamic criteria is a Ctrough level above 25 ug/ml in children and adolescents after the first subcutaneous dose.

SECONDARY OUTCOMES:
Number of participants achieving a repose of complete response (CR) | 1 year
  Response Evaluation Criteria in Solid Tumors (RECIST) criteria CR: complete disappearance of all target lesions.
Overall survival | 1 year
  Kaplan-Meier estimate
Progression-free survival | 1 year
  Kaplan-Meier estimate
Disease-free survival | 1 year
  Kaplan-Meier estimate

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Menon, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- UCI-Fred Hutch Cancer Centre, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menon MP, Ddungu H, Mubiru KR, Adams SV, Asea J, Namagembe R, Namuli P, Kambugu J, Towlerton AMH, Puronen C, Uldrick TS, Orem J, Warren EH. Phase I Study of Subcutaneous Rituximab Hyaluronidase Combined With CHOP Chemotherapy for the Treatment of Diffuse Large B-Cell Lymphoma in Uganda. JCO Glob Oncol. 2025 Apr;11:e2400489. doi: 10.1200/GO-24-00489. Epub 2025 Apr 4. PMID 40184567

DOCUMENTS (1):
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03864419/ICF_000.pdf